CLINICAL TRIAL: NCT01574118
Title: Enhancing Exposure Therapy for PTSD: An Investigation of Non-Pharmacological Augmentation Strategies
Brief Title: Enhancing Exposure Therapy for Post-traumatic Stress Disorder
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: COVID-19
Sponsor: University of Texas at Austin (Other)
Collaborators: University of Pennsylvania (Other)
Responsible Party: Principal Investigator, Michael J. Telch, Principal Investigator, University of Texas at Austin
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: 2012-02-0100
Record Dates: First submitted 2012-04-03; First posted 2012-04-10 (Estimated); Last update posted 2022-08-29 (Actual); Status verified 2022-08

CONDITIONS: Chronic Posttraumatic Stress Disorder
Keywords: PTSD; Posttraumatic Stress Disorder; Exposure Therapy; Prolonged Exposure; Fear Memory Retrieval; Compound extinction; Deepened extinction; Psychotherapy
MeSH Terms: conditions — Stress Disorders, Post-Traumatic

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Brief Enhanaced Exposure Therapy (Experimental): The following interventions are included in this arm:
  1. Psycho-education addressing common reactions to trauma
  2. Revisiting the Trauma memories
  3. Processing the trauma memories
  4. In vivo Exposure homework
  5. *Use of a brief pre-exposure trauma memory retrieval trial
  6. Exposure to video clips related to the patient's trauma
  7. Compound extinction - simultaneously exposing patient to trauma video clips while they listen to their trauma script
  Interventions: Behavioral: Revisiting the Trauma memories; Behavioral: Processing the trauma memories; Behavioral: Psychoeducation; Behavioral: Trauma Memory Retrieval Trial; Behavioral: Exposure to video clips related to the patient's trauma; Behavioral: Exposure Homework; Behavioral: Compound extinction
- Standard Prolonged Exposure Therapy (Active Comparator): The following interventions are included in this arm:
  1. Psycho-education addressing common reactions to trauma
  2. Revisiting of the Trauma memories
  3. Processing the trauma memories
  4. Breathing retraining
  5. In vivo Exposure homework
  Interventions: Behavioral: Revisiting the Trauma memories; Behavioral: Processing the trauma memories; Behavioral: Psychoeducation; Behavioral: Breathing retraining; Behavioral: Exposure Homework
- Delayed Treatment Control (No Intervention): Patients assigned to this arm receive assessment only (Week 0, 3, and 6) prior to receiving standard prolonged exposure therapy using the Foa et al treatment manual.

INTERVENTIONS:
Behavioral: Revisiting the Trauma memories — Patient engages in repeated revisiting of their trauma memory under the guidance of the therapist for about 40 minutes. During each revisiting trial the patient closes their eyes and verbally describes the trauma and the feeling and thoughts experienced during the trauma.
  Other Names: Trauma Revisiting
  Arms: Brief Enhanaced Exposure Therapy; Standard Prolonged Exposure Therapy
Behavioral: Processing the trauma memories — The patient and therapist discuss the patient's experience during the trauma revisiting with the goal of helping the patient gain alternative perspectives of the trauma.
  Other Names: Trauma Processing
  Arms: Brief Enhanaced Exposure Therapy; Standard Prolonged Exposure Therapy
Behavioral: Psychoeducation — Through patient handouts and didactic instruction, the patient learns about the common reactions to trauma and the rationale for exposure therapy.
  Arms: Brief Enhanaced Exposure Therapy; Standard Prolonged Exposure Therapy
Behavioral: Trauma Memory Retrieval Trial — Prior to the start of Imaginal Exposure, the patient is asked to recall a threatening element of their trauma memory for 1 minute. This is followed by a 30-minute rest-period prior to beginning imaginal exposure.
  Other Names: Fear Retrieval
  Arms: Brief Enhanaced Exposure Therapy
Behavioral: Exposure to video clips related to the patient's trauma — Patient is seated in front of a computer monitor and instructed to view a 30-min looped video clip that thematically resembles the patient's trauma.
  Other Names: Exposure to trauma clips
  Arms: Brief Enhanaced Exposure Therapy
Behavioral: Breathing retraining — Patient is seated comfortably in a chair and instructed to breathe slowly and deeply in a relaxed manner.
  Other Names: Relaxed breathing
  Arms: Standard Prolonged Exposure Therapy
Behavioral: Exposure Homework — Therapist assists the patient in identifying trauma-related situations/activities that the patient is avoiding and encourages the patient to begin to confront these situations between sessions.
  Other Names: In vivo exposure outside of session
  Arms: Brief Enhanaced Exposure Therapy; Standard Prolonged Exposure Therapy
Behavioral: Compound extinction — The patient repeatedly confronts the truama-related media clip while simultaneously listening to their own trauma script through headphones.
  Other Names: Deepened Extinction
  Arms: Brief Enhanaced Exposure Therapy

SUMMARY:
This study is investigating a new brief psychotherapy for post-traumatic stress disorder (PTSD) which, modifies an already proven psychotherapy for PTSD by adding two new components and modifying several others. The goal of the study is to determine whether this experimental treatment outperforms the well-established standard treatment.

DETAILED DESCRIPTION:
This study is investigating a new brief psychotherapy for post-traumatic stress disorder (PTSD) which, modifies an already proven psychotherapy for PTSD by adding two new components and modifying several others. The goal of the study is to determine whether this experimental treatment outperforms the well-established standard treatment. Individuals between the ages of 18-65 with chronic PTSD are randomly assigned to one of three psychotherapy conditions: (a) brief enhanced exposure therapy; (b) standard prolonged exposure therapy; and (c) delayed standard exposure therapy. All study participants undergo a phone and face-to-face screening assessment to determine study eligibility and baseline (pretreatment-Week 0) symptom severity. Upon completing treatment, participants undergo three additional assessment visits (Week 6, Week 10, and Week 22). During each of these outcome assessment visits, participants complete a structured clinical interview and a battery of computer-administered questionnaires.

ELIGIBILITY:
Inclusion Criteria:

1. Current primary PTSD diagnosis based on DSM-IV criteria, with a minimum duration of 12 weeks since the traumatic event.
2. Between the age of 18 and 65.
3. Medication status stable for at least 6 weeks

Exclusion Criteria:

1. Current diagnosis of schizophrenia, delusional disorder, or organic mental disorder as defined by the DSM-IV.
2. Current diagnosis of bipolar disorder, depression with psychotic features, or depression severe enough to require immediate psychiatric treatment (i.e., serious suicide risk with intent and plan).
3. Current diagnosis of alcohol or substance dependence within the 3 previous months.
4. Unwilling or unable to discontinue current trauma-focused psychotherapy.
5. Ongoing intimate relationship with the perpetrator (in assault-related PTSD cases).
6. Other severe acute or chronic medical or psychiatric condition that, in the judgment of the Medical Director, would make the participant inappropriate for entry.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2012-04; Primary Completion 2020-03 (Actual); Study Completion 2020-03 (Actual)

PRIMARY OUTCOMES:
Change from baseline in PTSD symptom severity | Weeks 6, 10, 22
  PTSD Symptom Scale - Interview Version

SECONDARY OUTCOMES:
Change from baseline in depression symptom severity | Weeks 6, 10, 22.
  Quick Inventory of Depressive Symptomatology - Self-Report
Change from baseline in trauma-related cognitions | Weeks 6, 10, 22.
  Post-Traumatic Cognitions Inventory - Self-Report
Change from baseline in general physical and psychological health | Weeks 6, 10, 22
  Medical Outcomes Study Short Form 36, Version 2 - Self-report
Change from baseline in work, social/leisure activities, and family/home life functioning | Weeks 6, 10, 22.
  Sheehan Disability Scale - Self-report

CONTACTS AND LOCATIONS:
Overall Officials: Michael J Telch, Ph.D., Principal Investigator — University of Texas at Austin
Locations (1):
- Laboratory for the Study of Anxiety Disorders, University of Texas at Austin, Austin, Texas, United States